CLINICAL TRIAL: NCT01988038
Title: Repository Study of Autosomal Dominant Polycystic Kidney Disease
Acronym: Repository
Status: Withdrawn | Type: Observational
Why Stopped: No participants were enrolled.
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1305013979
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Polycystic Kidney Disease; Autosomal Dominant Polycystic Kidney Disease; Disease Progression
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Blood sample for genotyping of specific PKD1 and PKD2 mutations. Buccal and/or semen sample (optional and only if needed)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The design and establishment of the Polycystic Kidney Disease (PKD) Data Repository does not require, and may be constrained by, a narrowly conceived hypothesis. However, the PKD Repository has been designed to include demographic, clinical, biochemical, and genetic data that will further explore the natural history of the disorder and assess the factors that are likely to be associated with the progression of disease and the incidence of complications including renal failure, cardiovascular disease, and stroke.

DETAILED DESCRIPTION:
The goal of this project is to collect data from a large population of patients with PKD. Based upon the estimated prevalence of PKD (1:500 and 1:1000 live births), it is estimated that there may be 10,000 PKD patients in the New York City area. This sample size far exceeds any database established thus far. As many as 40% of affected PKD patients are reportedly unaware of a family history of this disease, in part because many patients may go undiagnosed until they present with a medical complication (e.g., hypertension, kidney failure). Furthermore, this initiative will provide an opportunity to compare data from racially diverse populations.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18 years and older
* Previously diagnosed with ADPKD

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled in this study will have the diagnosis of autosomal dominant polycystic kidney disease (ADPKD). The diagnostic criteria for at-risk individuals (i.e., with a first degree family member with ADPKD) includes the presence of at least two (unilateral or bilateral) renal cysts, and two cysts in each kidney are considered sufficient for diagnosis in aged 15 to 29 years and in 30 to 59 years, respectively. In families of unknown genotype, the presence of one or more (unilateral or bilateral) renal cysts is sufficient for establishing the diagnosis in individuals aged 15 to 29 years, two or more cysts in each kidney is sufficient for individuals aged 30-49 years.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Natural history of Autosomal Dominant Polycystic Kidney Disease (ADPKD) progression | Up to 20 years
  The primary interest of this protocol is to characterize the renal and extrarenal manifestations of ADPKD, evaluate the natural history of the disease progression, and explore potential associations between PKD gene variants and ADPKD phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Blumenfeld, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States